## SIT Internal



## [Participant Consent Form]

| Project Title: | | Development of a novel Asian Mediterranean Diet and its acceptability in Non-Alcoholic Fatty Liver Disease (NAFLD) – a pre-intervention study.("Research") |
|---|---|---|
| SIT-IF | RB Application No.: | RECAS-0244 |
| Please | tick accordingly: | |
| | I voluntarily agree to tak | e part in this Research. |
| | Appendix 1). The invest and likely duration of the health information and/o | opy of the Participant Information Sheet for this Research (attached as igators have given me a full explanation on the nature, purpose, location Research, what I will be expected to do, as well as how my personal data r biological materials will be used. I have been given the opportunity to ask of this Research and have understood the advice and information given. |
| | without justifying my ounderstand that my with | free to withdraw my consent to participate in this Research at any time decision and without prejudice and consequence whatsoever. I also drawal of consent does not affect the research information obtained before and such information may be retained and used for this Research |
| | all personal data relating | e of my personal data for the purpose of this Research. I understand that<br>g to this Research is held and processed in the strictest confidence, and in<br>evant data protection laws in Singapore. |
| | I agree to be contacted | for matters relating to this Research. |
| | I agree to the photo-taking/ audio-recording/ video-recording of my participation in the Research. I understand and agree that although my name will be not associated with the photographs/ audio recording/ video-recordings used in publication/presentation, I may still be identified. | |
| | esearch has been explain<br>of consent taker). | ed to me in <u>English</u> , which I understand, by |
| Name a | and Signature (Participan | t) Date |
| Name a | and Signature (Consent 1 | Taker) Date |

Date

For further information on the above research study or to provide feedback, please contact:

- Verena Tan (Principal Investigator) <u>verena.tan@singaporeetech.edu.sg</u>
  Gary Chiah Tung Lin (Co-Investigator) <u>gary.chiah@singaporetech.edu.sg</u>

Name and Signature (Witness)